CLINICAL TRIAL: NCT04258163
Title: Association of Survival With Maintenance Therapy in Patients With Metastatic Breast Cancer After First-line Chemotherapy
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2019-099
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Maintenance Chemotherapy; Maintenance Endocrine Therapy; Overall Survival; Safety
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Maintenance Chemotherapy; liposomal doxorubicin; Gemcitabine; Fulvestrant; Anastrozole; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- MCT Group: People who received chemotherapy as a maintenance therapy after first-line chemotherapy reaching a state of no progress for at least 4 weeks. One patient only received one of the intervention drugs for maintenance therapy.
  Interventions: Drug: Capecitabine; Drug: Liposomal doxorubicin; Drug: Gemcitabine
- MET Group: People who received endocrine therapy as a maintenance therapy after first-line chemotherapy reaching a state of no progress for at least 4 weeks. One patient only received one of the intervention drugs for maintenance therapy.
  Interventions: Drug: Fulvestrant; Drug: Anastrozole; Drug: Letrozole
- Observation Group: People who didn't receive any maintenance therapy after first-line chemotherapy reaching a state of no progress for at least 4 weeks.

INTERVENTIONS:
Drug: Capecitabine — 1000-1250 mg/m 2 PO twice daily days 1-14, cycled every 28 days
  Other Names: Maintenance Chemotherapy
  Groups: MCT Group
Drug: Liposomal doxorubicin — 50 mg/m 2 IV day 1, cycled every 28 days
  Other Names: Maintenance Chemotherapy
  Groups: MCT Group
Drug: Gemcitabine — 800-1200 mg/m 2 IV days 1, 8, and 15, cycled every 28 days
  Other Names: Maintenance Chemotherapy
  Groups: MCT Group
Drug: Fulvestrant — 500mg IH Days 0, 14, 28, then every 28 days
  Other Names: Maintenance Endocrine Therapy
  Groups: MET Group
Drug: Anastrozole — 1mg PO qd
  Other Names: Maintenance Endocrine Therapy
  Groups: MET Group
Drug: Letrozole — 2.5mg PO qd
  Other Names: Maintenance Endocrine Therapy
  Groups: MET Group

SUMMARY:
To investigate the benefits and risks of maintenance chemotherapy (MCT), maintenance endocrine therapy (MET) and none maintenance therapy after first-line treatment of metastatic breast cancer (MBC).

DETAILED DESCRIPTION:
There are several options for MBC patients who are responding to chemotherapy, to continue treatment with a fix number of cycles or until disease progression which also known as maintenance chemotherapy (MCT), to stop chemotherapy and take a watch and wait strategy, or to stop chemotherapy and start the maintenance endocrine therapy (MET) for hormone receptor (HR) positive patients. Since the role of maintenance therapy in prolonging the overall survival (OS) and progression-free survival (PFS) of MBC was controversial in previous studies, the investigators performed a systematic review of randomized controlled trials to detect the association of survival with maintenance therapy in patients with MBC after first-line chemotherapy. And the investigators further performed a multi-center retrospective real-world study to evaluate these two maintenance modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically clear invasive breast cancer between 2003 and 2018;
* Female,18-75 years old;
* Measurable metastatic lesion according to RECIST 1.1 evaluation criteria;
* The first-line chemotherapy regimen is a breast cancer combination or single-agent chemotherapy regimen recommended by the NCCN guidelines;
* First-line chemotherapy is effective (according to RECIST1.1 evaluation criteria, the efficacy is evaluated as complete response (CR), partial response (PR), or steady state (SD));
* After the last cycle of first-line chemotherapy, patients should still be in a state of no progress for at least 4 weeks;
* Patients' Karnofsky performance status (KPS) scores were ≥70.

Exclusion Criteria:

* Unmeasurable metastatic lesion according to RECIST 1.1 evaluation criteria.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi-center real world study to compare maintenance chemotherapy (MCT), maintenance endocrine therapy (MET) and observation in patients with HR-positive MBC who achieved disease control after first-line chemotherapy. Patients were retrospectively enrolled from 3 different medical center.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Estimated 36 months
  From enrollment to death (for any reason)

SECONDARY OUTCOMES:
Progression free survival (PFS) | Estimated 18 months
  From enrollment to progression or death (for any reason)

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, PhD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (3):
- China (3):
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ren W, Yu Y, Hong H, Wang Y, Gao Q, Chen Y, Chen P, Zhao J, Ou Q, Lin D, Fu T, Tan Y, Li C, Xie X, Ye G, Tang J, Yao H. Clinical Evidence of Chemotherapy or Endocrine Therapy Maintenance in Patients with Metastatic Breast Cancer: Meta-Analysis of Randomized Clinical Trials and Propensity Score Matching of Multicenter Cohort Study. Cancer Res Treat. 2022 Oct;54(4):1038-1052. doi: 10.4143/crt.2021.698. Epub 2022 Feb 4. PMID 35130417